CLINICAL TRIAL: NCT04184050
Title: A Phase 1 Open-label, Multicenter, Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of HPN217 in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of HPN217 in Participants With Relapsed/Refractory Multiple Myeloma MK-4002 (MK-4002-001)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Harpoon Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HPN217-3001; U1111-1261-6031 (Registry Identifier: UTN); MK-4002-001 (Other: MSD); 2024-515582-33-00 (Registry Identifier: EU CT); 2019-004793-26 (EudraCT Number)
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma; Multiple Myeloma of Bone; Multiple Myeloma With Failed Remission
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-4002 monotherapy dose escalation (Experimental): MK-4002 is intravenously (IV) administered once weekly in escalating doses.
  Interventions: Drug: MK-4002
- MK-4002 dose escalation with extended dosing intervals (Experimental): MK-4002 is IV administered once every 2 weeks.
  Interventions: Drug: MK-4002

INTERVENTIONS:
Drug: MK-4002 — IV infusion
  Other Names: HPN217

SUMMARY:
Researchers want to learn if MK-4002 (also known as HPN217) can treat relapsed or refractory multiple myeloma (RRMM). The goals of this study are to learn about the safety of different doses of MK-4002 and how well people tolerate them. Researchers also want to learn what happens to different doses of MK-4002 in a person's body over time.

ELIGIBILITY:
Major Inclusion Criteria:

1. Patients ≥18 years of age at the time of signing informed consent
2. Documented RRMM for which no standard therapy options are anticipated to result in a durable remission. Relapse defined as progressive disease after initial response (minimal response [MR] or better) to previous treatment, more than 60 days after cessation of last treatment. Refractory disease defined as <25% reduction in M protein or progression of disease during treatment or within 60 days after cessation of treatment.
3. Received at least 3 prior therapies (including proteasome inhibitor, immune modulatory drug, and an anti-CD38 antibody; patients should not be a candidate for or be intolerant of all established therapies known to provide clinical benefit in multiple myeloma).
4. Measurable disease defined as at least one of the following:

   1. Serum M-protein ≥0.5 g/dL
   2. Urine M-protein ≥200 mg/24 hours
   3. Serum free light chain (FLC) assay: Involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
5. Resolved acute effects of any prior therapy to baseline severity or Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade ≤1.

Major Exclusion Criteria:

1. Plasma cell leukemia; non-secretory myeloma (e.g., solitary plasmacytoma)
2. Patients with only extramedullary relapse of multiple myeloma who do not meet requirement for measurable disease.
3. Prior autologous peripheral stem cell transplant or prior autologous bone marrow transplantation within <90 days of the start of study
4. Prior allogeneic stem cell transplantation or solid organ transplantation within 12 months of Screening. However, any patient receiving immunosuppressive medication will be excluded.
5. History of or known or suspected autoimmune disease (exception(s): patients with vitiligo, resolved childhood atopic dermatitis, hypothyroidism, or hyperthyroidism that is clinically euthyroid at Screening are allowed). Other exceptions may be allowed following discussion with the Sponsor Medical Monitor for patients who have not received any treatment for their autoimmune disorder in the past 3 years
6. Second primary malignancy that has not been in remission for greater than 3 years. Exceptions that do not require a 3-year remission: non-melanoma skin cancer, resected melanoma in situ, in situ cervical cancer, adequately treated Stage I cancer from which the subject is currently in remission and has been in remission for ≥2 years, low-risk prostate cancer with Gleason score <7 and prostate-specific antigen <10 ng/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to ~6 years
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. A TEAE is an adverse event that occurs on or after the first dose of study treatment. The number of participants with TEAEs graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (American Society for Transplant and Cellular Therapy [ASTCT] grading criteria for cytokine release syndrome [CRS] and immune effector cell-associated neurotoxicity syndrome [ICANS]) will be reported.
Number of Participants Who Discontinued Study Treatment Due to an AE | Up to ~6 years
  An AE is defined as any untoward medical occurrence in a participant administered study drug, which does not necessarily have to have a causal relationship with the study drug. The number of participants who discontinue study treatment due to an AE will be reported.
Number of Participants with Dose-limiting toxicities (DLT) | Up to 35 days in Cycle 1
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the CTCAE 5.0 version for all AEs except CRS and ICANS, which will be graded according to ASTCT. The number of participants who experience a DLT will be reported.
Single Dose Maximum Serum Concentration (Cmax) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the Cmax of MK-4002 after a single dose.
Single Dose Time to Maximum Concentration (Tmax) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the Tmax of MK-4002 after a single dose.
Area Under the Single Dose Concentration-time Curve Over the Dosing Interval τ (AUCsd,τ) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the AUCsd,τ of MK-4002.
Single Dose Area Under the Concentration-time Curve Extrapolated to Infinity (AUCinf) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the AUCinf after a single dose of MK-4002.
Single Dose Terminal Elimination Half-life (t1/2) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the t1/2 after a single dose of MK-4002.
Single Dose Clearance (CL) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the CL after a single dose of MK-4002.
Multiple Dose Maximum Concentration at Steady State (Css,max) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the Css,max of MK-4002. This outcome will be analyzed only if steady state is achieved, and data are available.
Multiple Dose Time to Maximum Concentration at Steady State (Tss,max) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the Tss,max of MK-4002. This outcome will be analyzed only if steady state is achieved, and data are available.
Mutiple Dose Area Under the Steady State Concentration-time Curve Over the Dosing Interval τ (AUCss,τ) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the (AUCss,τ) of MK-4002. This outcome will be analyzed only if steady state is achieved, and data are available.
Multiple Dose Terminal Elimination Half-life (t1/2) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the t1/2 of MK-4002. This outcome will be analyzed only if steady state is achieved, and data are available.
Multiple Dose Minimum Concentration at Steady State (Css,min) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the Css,min of MK-4002. This outcome will be analyzed only if steady state is achieved, and data are available.
Multiple Dose Clearance (CL) | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the CL of MK-4002. This outcome will be analyzed only if steady state is achieved, and data are available.
Multiple Dose Volume of Distribution at Steady State (Vss) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the Vss of MK-4002. This outcome will be analyzed only if steady state is achieved, and data are available.
Multiple Dose Accumulation Ratio (AUCss,τ/AUCsd,τ) of MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the (AUCss,τ/AUCsd,τ) of MK-4002. This outcome will be analyzed only if steady state is achieved, and data are available.

SECONDARY OUTCOMES:
Best Overall Response Rate (BOR) | Up to ~6 years
  BOR is defined as the participant's best disease response assessed during the study. BOR will be based on assessments collected after the first dose of study drug until disease progression is documented.
Overall Response rate (ORR) | Up to ~6 years
  ORR is defined as the percentage of the participants with either a stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) according to the International Myeloma Working Group (IMWG) Response Criteria. CR = negative immunofixation of serum and urine AND <5% plasma cells in the bone marrow; sCR = CR plus normal serum free light-chain (FLC) assay ratio and absence of clonal plasma cells in bone marrow; VGPR = serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein plus urine M-protein <100 mg/24 hr; PR = ≥50% reduction of serum M- protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. The percentage of participants who experience CR or PR will be presented.
Progression-free Survival (PFS) | Up to ~6 years
  PFS is defined as the time from first dose of study drug to documented disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to ~6 years
  OS is defined as the time from first dose of study drug to death due to any cause.
Duration of Response (DOR) | Up to ~6 years
  DOR is defined as the time from the first observed response observed response (sCR, CR, VGPR, or PR) to documented disease progression or death due to any cause. CR = negative immunofixation of serum and urine AND <5% plasma cells in the bone marrow; sCR = CR plus normal serum free light-chain (FLC) assay ratio and absence of clonal plasma cells in bone marrow; VGPR = serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein plus urine M-protein <100 mg/24 hr; PR = ≥50% reduction of serum M- protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. DOR as assessed by investigator according to IMWG response criteria will be presented.
Time to Response (TTR) | Up to ~6 years
  TTR is defined as the time from first dose of study drug to the first observed response response (sCR, CR, VGPR, or PR). CR = negative immunofixation of serum and urine AND <5% plasma cells in the bone marrow; sCR = CR plus normal serum free light-chain (FLC) assay ratio and absence of clonal plasma cells in bone marrow; VGPR = serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein plus urine M-protein <100 mg/24 hr; PR = ≥50% reduction of serum M- protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. TTR as assessed by investigator according to IMWG response criteria will be presented.
Number of Participants with Anti-drug Antibodies (ADAs) against MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the ADA response against MK-4002. The number of ADAs will be presented.
Titers of ADAs against MK-4002 | At designated timepoints (up to ~6 years)
  Blood samples collected at designated time points will be used to determine the titers of ADAs against MK-4002.
Percentage of Participants Who are Minimal Residual Disease (MRD) Negative | At designated timepoints (up to ~6 years)
  Bone marrow samples will be used to determine the MRD negative. MRD is defined as the percentage of patients who achieve an sCR or CR who meet MRD Criteria for Sequencing MRD-negative rate at 10^5 nucleated cells threshold and at 10^6 nucleated cells threshold. CR = negative immunofixation of serum and urine AND <5% plasma cells in the bone marrow; sCR = stringent complete response. Sequencing MRD-negative is the absence of clonal plasma cells by next-generation sequencing (NGS) on bone marrow aspirate in which presence of a clone is defined as less than 2 identical sequencing reads obtained after deoxyribonucleic acid (DNA) sequencing of bone marrow aspirates using the LymphoSIGHT platform (or validated equivalent method).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (12):
- United States (8):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The University of Kansas Cancer Center, Fairway, Kansas
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University of Rochester James P Wilmot Cancer Institute, Rochester, New York
  - OHSU, Portland, Oregon
  - University of Washington - Seattle Cancer Center Alliance, Seattle, Washington
- France (2):
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
- Spain (2):
  - Josep Carreras Leukaemia Research Institute, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz (UAM-FJD), Madrid

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26141&tenant=MT_MSD_9011